CLINICAL TRIAL: NCT06053775
Title: Intervention With Non-Invasive Brain Stimulation and Cognitive Training for Depressive Symptomatology Associated With Breast Cancer (ONCODEP)
Brief Title: Non-Invasive Brain Stimulation and Cognitive Training for Depressive Symptomatology Related to Breast Cancer (ONCODEP)
Acronym: ONCODEP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Collaborators: Fundacin Biomedica Galicia Sur (Other)
Responsible Party: Principal Investigator, María Teresa Carrillo de la Peña, University Professor, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023/213; FPU21/00082 (Other Grant/Funding Number: Ayudas para contratos predoctorales FPU 2021)
Record Dates: First submitted 2023-09-11; First posted 2023-09-26 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Depressive Symptoms; Cognitive Impairment
Keywords: Non-Invasive Brain Stimulation; Cognitive Training; Depressive Symptoms; Cognitve Impairment; Breast Cancer
MeSH Terms: conditions — Depression; Cognitive Dysfunction; Breast Neoplasms | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized, four-arm, placebo-controlled, parallel-structured, double-blinded clinical trial.
Who Masked: Participant, Investigator
Masking Description: In this study, a double-blind design will be used, since the device used for the tDCS/tACS intervention allows for total blinding. The patient and the researchers involved in treatment will be blinded to the group of treatment (except for the OCT group). Evaluation and data analysis will be blinded to group assignment until the participant has completed the study. Only the members of the research team in charge of generating the randomization list will have access to the patient's intervention status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Online Cognitive Training (Active Comparator): 15 sessions of 20 minutes each one.Training will focus on the stimulation of several cognitive functions (attention, memory and learning, language, executive functions,processing speed, etc) through different exercises. The sessions will be adjusted to the individual performance level. The participant will perform these exercises from their computer or tablet, through the NeuronUp2GO platform, and the researcher will have access to all the session data.
  Interventions: Device: Online Cognitive Training
- Transcranial Direct Current Stimulation (Experimental): tDCS: 15 daily sessions targeting left DLPFC (anode: F3, cathode: Fp2) Current intensity will be set at 2mA and will be applied for 20 minutes, with 15-second ramps up and down at the beginning and end of the stimulation period.
  During the session, the participant will be performing the OCT.
  Interventions: Device: Transcranial Direct Current Stimulation; Device: Online Cognitive Training
- Transcranial Alternating Current Stimulation (Experimental): tACS: 15 daily sessions targeting left DLPFC (anodes: F3, F4; frequency: 4Hz -theta-tACS-). Current intensity will be set at 2mA and will be applied for 20 minutes, with 15-second ramps up and down at the beginning and end of the stimulation period.
  Participant will be performing the OCT during stimulation.
  Interventions: Device: Transcranial Alternating Current Stimulation; Device: Online Cognitive Training
- tES sham (Sham Comparator): 15 sessions of sham stimulation for 20 minutes, acting as a placebo control group. The electrode montage will be the same as that used in the active neuromodulation conditions: tDCS for half of the participants and tACS for the other half. In this sham stimulation condition, the current will only be delivered for a 15 seconds, at the ramp-up and ramp-down times at the beginning and end of the session.
  The OCT will also be the same as those performed by participants in the other groups
  Interventions: Device: tES sham; Device: Online Cognitive Training

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — tDCS+OCT
  Other Names: tDCS
  Arms: Transcranial Direct Current Stimulation
Device: Transcranial Alternating Current Stimulation — tACS+OCT
  Other Names: tACS
  Arms: Transcranial Alternating Current Stimulation
Device: tES sham — tES sham + OCT
  Arms: tES sham
Device: Online Cognitive Training — OCT
  Other Names: OCT

SUMMARY:
The goal of this clinical trial is to test a home-delivered intervention that combines Non-Invasive Brain Stimulation techniques (transcranial direct and alternating current stimulation -tDCS and tACS-) and Online Cognitive Training (OCT) to treat depressive symptomatology and cognitive decline associated with breast cancer. The main questions aims to be answered are:

* To analyze the efficacy and feasibility of the intervention to treat depressive symptomatology.
* To analyze the efficacy and feasibility of the intervention to treat cognitive decline.
* To evaluate the medium and long-term effects (1, 3 and 6 months) of intervention.

An OCT program and a portable wireless tDCS/tACS system will be used to perform the intervention at home. Patients will be divided into four treatment groups, depending on whether they will receive the OCT applied independently or combined with tDCS/tACS active or sham.

In addition, saliva samples will be collected to identify bomarkers predictive of treatment efficacy.

DETAILED DESCRIPTION:
This study is aimed at analyzing the feasibility and therapeutic efficacy of a home-based treatment using tDCS/tACS and an OCT program to treat depressive symptomatology (primary outcome variable) associated with breast cancer.The effect of the intervention on the patients' cognitive functioning (secondary outcome variable) will be also studied. In addition, saliva biomarkers and other clinical variables will be analyzed to determine whether they are related to the response to treatment. Finally, the impact of the intervention on the burden of the relatives/caregivers will be studied.

Oncology Units of the Galician Health Service will be contacted for recruitment. Oncologists will review whether patients meet the inclusion criteria and none of the exclusion criteria. If so, patients will be given an information flyer and will contact the research team to receive more information and, if they wish, to participate in the study. If patients are interested in participating, researchers will contact them to confirm the inclusion/exclusion criteria and participants will be invited to the first face-to-face session. In this session, informed consent will be signed, pre-treatment neuropsychological assessment will be performed, medical data will be reviewed, and a saliva sample will be collected. After collecting this data, the first treatment session will take place in the presence of the researcher. The type of treatment each patient will receive (OCT, tDCS active+ OCT, tACS active+ OCT or sham neurostimulation+ OCT. ) will be chosen randomly, using a randomization list.

After that, each patient will undergo 14 sessions, daily, at home. The tES devices (Soterix Medical Inc) have been designed for home use and allow the application of the stimulation by the patient himself, while being monitored by the researcher. The OCT will be delivered through NeuronUp2GO platform.Possible adverse effects associated with neurostimulation (which are mild and transitory) and other variables that may affect its efficacy (medication diary, caffeine intake...) will be monitored daily.

Finally, a post-treatment assessment will be carried out 15 days after the start of treatment and a follow-up assessment will be carried out 1, 3 and 6 months after the end of treatment. The 15-day and 1 month assessments will be the same as the pre-treatment (questionnaries and neuropsychological test). The follow-ups at 3 and 6 months will be done online, by filling in questionnaires.

Both the treatment administration and analysis of the results will be blinded.

First, descriptive analyses will be performed on the sociodemographic and clinical data. To evaluate the efficacy of the treatments on depressive symptomatology and cognitive function, linear mixed models will be carried out. The dependent variable will be the test score, and treatment group, time (pre, post, follow-ups) and group*time interaction as fixed factors, and participants as random effects.

The possible modulating effect of sociodemograpchic and clinical variables on treatment efficacy will be analyzed. Also, for the clinical validation of the treatments, the analysis of the Minimal Clinically Important Difference (MCID) at short (15 days), medium (1 month) and long term (3 and 6 months) will be included. The difference between the pre- and post-treatment assessment in the primary and secondary variable scores should be equal to or greater than 30%.

Proteomic analysis will be performed at the Fundación Biomédica Galicia Sur. The following analysis will be performed: determination of total protein, mass spectrometry and electrophoretic separation of the samples by SDS-PAGE and identification of the bands of interest by Shotgun. The whole sample will be analyzed in liquid mass spectrometer (LC-MS/MS). Linear or logistic regression analysis will be performed to determine the predictive power of the saliva biomarkerson treatment efficacy.

Since the present research involves adult humans, it will be conducted under applicable international, EU and national laws and regulations (The Declaration of Helsinki: Ethical Principles for Medical Research Involving Human Subjects; The International Conference on Harmonisation (ICH)/Good Clinical Practice (GCP) Guidelines; the Convention for the Protection of Human Rights and Dignity of the Human Being with regard to the Application of Biology and Medicine; and the UNESCO Universal Declaration on Bioethics and Human Rights (2005). Permission has been obtained from the local IRB committee (CEIm de Galicia) to conduct the study.

In terms of data protection, this study complies with the directives of the General Data Protection Regulation (GDPR), approved by the European Commission on April 27, 2016 (EU 2016/679) and with the Organic Law 3/2018, of December 5, 2018, on the Protection of Personal Data and guarantees of digital rights. The storage and treatment of the samples will be carried out in accordance with the Biomedical Research Law 14/2007 and RD 1716/201.

Patients' clinical data will be collected in the study-specific data collection notebook using REDCap (Research Electronic Data Capture), a secure web-based application for building and managing online surveys and databases. Data collection will be pseudo-anonymous, protecting the identity of the participant. Only the principal investigator of the entity responsible for data collection (USC) will know the pseudonymization codes. The research team will have access to all coded data collected for the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer in early stages (life expectancy greater than 12 months).
* Patients who are receiving or have finished (maximum 6 months prior to participation in the participating in the study) some type of oncological treatment (Chemotherapy, Radiotherapy, Immunotherapy, Hormonal Therapy).
* Patients whose mother tongue is Galician or Spanish.
* Ability to give informed consent.
* Present depressive symptomatology: score of 4 or higher in the BDI-FS.
* Ability to use WhastApp
* Have access to some technology (desktop computer, laptop or tablet) and the Internet (Firefox or Chrome browsers).

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Patients with metastasis.
* Patients with a mental health disorder (major depressive disorder, bipolar,anxious, psychotic...) diagnosed by a psychiatrist prior to the oncological process.
* Patients with a history of cognitive impairment or dementia prior to the oncologic process.

oncological process.

* Patients with a history of neurosurgery, cortical lesions or neurological alterations prior to the oncological process.
* Patients with history or current consumption of non-prescribed drugs.
* Patients with the following medication regimen: mood stabilizers, antipsychotics, anticonvulsants, l-dopa, rivastigmine, dextromethorphan, flunarizine, sulpiride, use of benzodiazepines (excluding long half-life benzodiazepines (Bromazepam, Diazepam) on a continuous/habitual basis,Alprazolam >1mg per day, Lorazepam >2mg per day).
* Patients taking antidepressant medication should have a stable regimen ( same medication at the same dose for a minimum of four weeks prior to entering the study.The regimen with antidepressant drugs or drugs used as treatment to improve cognition should be kept stable during the entire participation (until the follow-up evaluation has been performed).
* Patients unable to complete a neuropsychological examination.
* Patients who are participating in a research study/clinical trial with drugs.
* Patients who present any condition contraindicated to undergo tES (intracranial ferromagnetic devices or implanted stimulators; history of active epilepsy; history of neurosurgery, traumatic brain injury with loss of brainwith loss of consciousness and/or cortical lesion) (Antal et al., 2017)

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory- Fast Screen (BDI-FS) | pre-, post- intervention (15 days) and follow-up (1,3,6 months)
  Screening of depressive symptoms in medical patients (7 items, scored on a Likert scale from 0 to 3). BDI-FS minimum and maximum values range from 0 to 21, with higher scores meaning more depressive symptomatology.

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS) Cognitive Function 8a | pre-, post- intervention (15 days) and follow-up (1,3,6 months)
  To assess subjective cognitive complaints in the last week (8 items, scored on a Likert scale from 1 to 5). Minimum and maximum values rang from 8 to 40. Lower scores mean more subjective cognitive complaints.
Montreal Cognitive Assessment (MoCA) | pre-, post- intervention (15 days) and follow-up (1month).
  Cognitive impairment screening that explores attention, concentration, executive functions, memory, language, visual-constructive abilities, calculation and orientation (10 minutes). Minimum and maximum values range from 0 to 30. Lower scores mean better cognitive functioning, The cutoff point for Mild Cognitive Impairment is 26.

OTHER OUTCOMES:
Digit Span Test (forward and backward) (Barcelona Test-Revised) | pre-, post- intervention (15 days) and follow up (1 month)
  To assess the verbal span and working memory with series of digits in increasing and decreasing order (5 minutes).
Spain-Complutense Verbal Learning Test (TAVEC) | pre-, follow-up (1 month)
  To examine recent and delayed verbal learning and memory delayed (30 minutes,including the delay between trials).
Verbal fluency test (NEURONORMA Project) | pre-, post- intervention (15 days) and follow up (1 month)
  To assess lexical and semantic fluency and executive components of language (5 minutes).
Salthouse Perceptual Comparison Test (SPCT) | pre-, post- intervention (15 days) and follow up (1 month)
  To examine perceptual comparison and processing speed (3 minutes).
Dual task | pre-, post- intervention (15 days) and follow up (1 month)
  Evaluate the response cost of performing a task individually or while performing it simultaneously. The tasks consist of recalling a series of digits in direct order and letter and symbol cancellation tasks.(5 minutes).
d2-R (Test of Attention-Revised) | pre-, post- intervention (15 days) and follow up (1 month)
  To assess examines selective attention and concentration using a cancellation task (10 minutes)
Generalized Anxiety Disorder-7 scale (GAD-7) | pre-, post- intervention (15 days) and follow-up (1 month)
  To assess anxious symptomatology (7 items, scored on a Likert scale from 0 to 3). Scores range between 0 and 21, with higher scores indicating higher anxious symptomatology.
PROMIS Fatigue 7a | pre-, post- intervention ( 15 days) and follow-up (1 month)
  To examine presence of fatigue symptoms (7 items, scored on a Likert scale from 1 to 5). Scores range between 7 and 35, with lower scores indicating higher fatigue symptoms.
EORTC QLQ-C30 | pre-, post- intervention (15 days) and follow-up (1,3,6 months)
  The QLQ-C30 is composed of both multi-item scales and single-item measures. The questionnaire icludes five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting), a global health status / QoL scale, and a number of single items assessing additional symptoms commonly reported by cancer patients.
  All of the scales and single-item measures range in score from 0 to 100.
  A high scale score represents a higher response level:
  * A high score for a functional scale represents a high / healthy level of functioning,
  * A high score for the global health status / QoL represents a high QoL,
  * A high score for a symptom scale / item represents a high level of symptomatology / problems.
Pittsburgh Sleep Quality Index (PSQI) | pre-, post- intervention (15 days) and follow-up (1 month)
  To assess sleep quality and disturbances over a 1-month. The questionnaire includes 19 items, combined to form seven scales to evaluate different components of sleep (subjective quality, latency, duration, efficiency, disturbances, medication use, sleep dysfunction). Each scale obtain a score that ranges from 0 to 3 (0- no difficulty, 3- severe difficulty). The 7 components are summed to obtain an overall quality o sleep score, from 0 to 21 points (0 - no difficulty, 21 - severe difficulty).
Zarit (Caregiver Burden Interview) | pre-, post- intervention (15 days) and follow-up (1,3,6 months)
  To assess the burden (stress and negative feelings) associated with the caregiving task. It is composed of 22 items answered according to a Likert scale range from 0 to 4. The cut-off point for caregiver burden is 46-47.
  It also makes a distinction between mild burden (up to 56) and heavy burden (more than 56).
Pain: ad-hoc questionnaire | pre-, post- intervention (15 days) and follow-up (1 month)
  It measures the change in pain intensity, interference and discomfort afeter the treatment. There are three scales (intensity, interference, discomfort), which score range from 1 (no pain, no interference, no discomfort) to 10 (unbearable pain, interferes greatly and very unpleasant). Lower scores indicate a lower presence of pain symptoms.
Self-efficacy: ad-hoc questionnaire | pre-, post- intervention (15 days) and follow-up ( 1 month)
  To analyze general and cognitive self-efficacy. 7 items scored on a Likert scale from 1 to 5. A higher score reflects greater confidence in achieving certain self-efficacy related goals.
Global improvement assessment: ad-hoc questionnaire | post- intervention (15 days) and follow-up (1, 3, 6 months)
  To know the subjective perception of improvement after treatment in terms of cognitive functioning, mood, fatigue, quality of sleep and quality of life. Each question is answered on a scale from 1 (no improvement) to 10 (great improvement).

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - University of Santiago de Compostela, Santiago de Compostela, A Coruña
  - Fundación Biomédica Galicia Sur, Vigo, Pontevedra

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lefaucheur JP, Antal A, Ayache SS, Benninger DH, Brunelin J, Cogiamanian F, Cotelli M, De Ridder D, Ferrucci R, Langguth B, Marangolo P, Mylius V, Nitsche MA, Padberg F, Palm U, Poulet E, Priori A, Rossi S, Schecklmann M, Vanneste S, Ziemann U, Garcia-Larrea L, Paulus W. Evidence-based guidelines on the therapeutic use of transcranial direct current stimulation (tDCS). Clin Neurophysiol. 2017 Jan;128(1):56-92. doi: 10.1016/j.clinph.2016.10.087. Epub 2016 Oct 29. PMID 27866120
- [Background] Moffa AH, Martin D, Alonzo A, Bennabi D, Blumberger DM, Bensenor IM, Daskalakis Z, Fregni F, Haffen E, Lisanby SH, Padberg F, Palm U, Razza LB, Sampaio-Jr B, Loo C, Brunoni AR. Efficacy and acceptability of transcranial direct current stimulation (tDCS) for major depressive disorder: An individual patient data meta-analysis. Prog Neuropsychopharmacol Biol Psychiatry. 2020 Apr 20;99:109836. doi: 10.1016/j.pnpbp.2019.109836. Epub 2019 Dec 16. PMID 31837388
- [Background] Rodella C, Bernini S, Panzarasa S, Sinforiani E, Picascia M, Quaglini S, Cavallini E, Vecchi T, Tassorelli C, Bottiroli S. A double-blind randomized controlled trial combining cognitive training (CoRe) and neurostimulation (tDCS) in the early stages of cognitive impairment. Aging Clin Exp Res. 2022 Jan;34(1):73-83. doi: 10.1007/s40520-021-01912-0. Epub 2021 Jun 22. PMID 34156651
- [Background] Cheng ASK, Wang X, Niu N, Liang M, Zeng Y. Neuropsychological Interventions for Cancer-Related Cognitive Impairment: A Network Meta-Analysis of Randomized Controlled Trials. Neuropsychol Rev. 2022 Dec;32(4):893-905. doi: 10.1007/s11065-021-09532-1. Epub 2022 Jan 29. PMID 35091967
- [Background] Gaynor AM, Pergolizzi D, Alici Y, Ryan E, McNeal K, Ahles TA, Root JC. Impact of transcranial direct current stimulation on sustained attention in breast cancer survivors: Evidence for feasibility, tolerability, and initial efficacy. Brain Stimul. 2020 Jul-Aug;13(4):1108-1116. doi: 10.1016/j.brs.2020.04.013. Epub 2020 Apr 27. PMID 32353419
- See also: tACS for the treatment of MDD — https://www.nature.com/articles/s41398-019-0439-0